CLINICAL TRIAL: NCT06300489
Title: Genotype-driven Phase I Study of Weekly Irinotecan Liposomes in Combination With Capecitabine-based Neoadjuvant Chemoradiation for Locally Advanced Rectal Cancer
Brief Title: Genotype-driven Weekly Irinotecan Liposomes in Combination With Capecitabine-based Neoadjuvant Chemoradiation for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARTOnG-2401
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- irinotecan liposomes+capecitabine+chemoradiotherapy (Experimental): There are three dose groups inciuding wild-type (GG+6/6)，unit site mutant (GG+6/7 or GA+6/6) and double sites mutant (GG+7/7 or AA+6/6 or GA+6/7)。Every group will receive irinotecan liposomes injection and capecitabine based chemoradiotherapy.
  Interventions: Drug: irinotecan liposomes+capecitabine

INTERVENTIONS:
Drug: irinotecan liposomes+capecitabine — Radiotherapy：IMRT DT 50Gy/25Fx. Capecitabine: 625mg/m2 bid po d1-5 qw. For patients are double sites mutant (GG+7/7 or AA+6/6 or GA+6/7)，the intial dose of Irinotecan liposomes is 25mg/m2 weekly，for four weeks。 This study stratify cases by the "3+3" rule according to UGT1A1 * 6 and UGT1A1 * 28 phenotypes. Three cases were enrolled in each dose group, and if there was no DLT, they were promoted to the next dose group（an increase of 5mg/m2）; If there is 1 case of DLT, 3 cases will be reenrolled in the same dose group. If there is no new occurrence of DLT, it will be promoted to the next dose group. Otherwise, the study will be terminated; If there are 2 cases of DLT, the study will be terminated, and the previous dose group will be the maximum tolerated dose (MTD).
  Other Names: chemoradiotherapy

SUMMARY:
This study is a multicenter, open, and phase I dose increasing clinical study. Based on the UGT1A1 * 28 and * 6 genotypes of patients with locally advanced rectal cancer, determine the dose limiting toxicity (DLT) and maximum tolerable dose (MTD) of weekly irinotecan liposomes in concurrent chemoradiotherapy with capecitabine, investigate the tolerance of irinotecan liposome combined with capecitabine in concurrent chemoradiotherapy with locally advanced rectal cancer, and recommend the dosage for Phase II clinical study，and explore the pharmacokinetic characteristics of irinotecan liposomes combined with capecitabine.At the same time，Preliminary observe the efficacy and safety of irinotecan liposomes combined with capecitabine in chemoradiotherapy.The study plans to recruit 30 patients with advanced rectal cancer who have not received any therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as rectal adenocarcinoma by histopathology, immunohistochemical pMMR or MSI-L, MSS;
2. The baseline clinical stage is T2-4 and/or N+, which is not suitable for initial local resection to achieve curative effect;
3. The distance between the tumor and the anus is<=10cm;
4. No distant metastasis;
5. Age range from 18 to 70 years old, regardless of gender;
6. ECOG PS score 0-1 points;
7. The UGT1A1 * 6 and UGT1A1 * 28 gene phenotypes are all wild-type (GG+6/6), unit point mutant (GG+6/7 or GA+6/6), and dual site mutant (GG+7/7 or AA+6/6 or GA+6/7);
8. Not receiving chemotherapy or any other anti-tumor treatment before enrollment;
9. Able to comply with the protocol during the research period;
10. Sign written informed consent.

Exclusion Criteria:

1. Diagnosed as rectal adenocarcinoma by pathological histology, and immunohistochemical dMMR or MSI-H;
2. UGT1A1 * 6, UGT1A1 * 28 gene phenotype three site mutations (AA+7/7 or AA+6/7 or GA+7/7);
3. Pregnant or lactating women
4. Individuals with a history of other malignant diseases in the past 5 years, excluding cured skin cancer and cervical cancer in situ
5. Individuals with a history of uncontrolled epilepsy, central nervous system disease, or mental disorders, whose clinical severity may be assessed by the researcher as hindering the signing of informed consent forms or affecting the patient's adherence to oral medication
6. Clinically severe (i.e. active) heart disease, such as symptomatic coronary heart disease, NYHA grade II or more severe congestive heart failure, or severe arrhythmia requiring medication intervention (see Appendix 12), or a history of myocardial infarction within the past 12 months
7. Organ transplantation requires immunosuppressive therapy
8. Severe uncontrolled recurrent infections or other serious uncontrolled comorbidities
9. The baseline blood routine and biochemical indicators of the subjects do not meet the following criteria: hemoglobin ≥ 90g/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; ALT and AST ≤ 2.5 times the normal upper limit value; ALP ≤ 2.5 times the normal upper limit value; Serum total bilirubin<1.5 times the upper normal limit value; Serum creatinine<1 times the upper normal limit value; Serum albumin ≥ 30g/L
10. Known individuals with dihydropyrimidine dehydrogenase (DPD) deficiency
11. Individuals who are allergic to any research medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-03 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
DLT（dose-limiting toxicity） | up to 6 months
  Any adverse event that occurs during a research period and is related to Irinotecan liposomes the and meets a certain level or higher of CTCAE.
MTD（maximum tolerable dose） | up to 6 months
  the highest dose of exposure to a substance without causing serious toxic reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No